CLINICAL TRIAL: NCT02852629
Title: Assessment of a Tool for Decision Making in Case of Worsening Condition of Cancer Patients
Acronym: CBP-Aggrav
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: CBP-AGGRAV_CIC
Record Dates: First submitted 2016-02-15; First posted 2016-08-02 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Lung Cancer
Keywords: decision-support sheet
MeSH Terms: conditions — Lung Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: observational study

SUMMARY:
Observational two year study to evaluate the utility of a decision-support sheet on how to proceed in case of aggravation of a patient's condition with advanced disease.

DETAILED DESCRIPTION:
Prospective and multicenter study conducted in the Rhône-Alpes-Auvergne area. All patients suffering from lung cancer admitted to a pulmonology unit in 2014 will be included. This document will be used if a decision to withhold life-sustaining treatment is decided. Investigators will assess the relationship between the planned intensity of care and those established when the patient develops an organ failure. Patient characteristics and factors associated with proposed levels and types of care will be analyzed. Patient and family opinions will be obtained after 3 months. The number of subjects is 468.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with lung cancer, hospitalized in pulmonology unit in one of the participating centers.
* Patient who requires a decision to withhold life-sustaining treatment
* One patient can be included at each hospitalization.

Exclusion Criteria:

* Minor patient
* Refusal of participation of the patient in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients will be recruited in the appreciation of the doctor (Md) of the service
Sampling Method: Non-Probability Sample
Enrollment: 483 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Emergent Serious Adverse Events | 1 year and a half
  The main objective of this study is to assess the relationship between the planned intensity of care and those established when the patient develops organ failure. The agreement will be assessed using Cohen's kappa coefficient .

SECONDARY OUTCOMES:
Patient feeling assessment using phone interview questionnaire | 3 months after patient inclusion
  Patients will be contacted by the investigator, to evaluate their feeling according to the collect of their opinion and wishes using a phone interview questionnaire within 30 minutes duration
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | first day
  assessment at inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toffart AC, Sakhri L, Girard N, Couraud S, Merle P, Fournel P, Perol M, Souquet PJ, Timsit JF, Moro-Sibilot D. [Assessment of a tool for decision making in case of worsening condition of cancer patients]. Rev Mal Respir. 2015 Jan;32(1):66-72. doi: 10.1016/j.rmr.2014.02.006. Epub 2014 Mar 20. French. PMID 25618207
- [Background] Toffart AC, Pizarro CA, Schwebel C, Sakhri L, Minet C, Duruisseaux M, Azoulay E, Moro-Sibilot D, Timsit JF. Selection criteria for intensive care unit referral of lung cancer patients: a pilot study. Eur Respir J. 2015 Feb;45(2):491-500. doi: 10.1183/09031936.00118114. Epub 2014 Oct 16. PMID 25323247
- [Background] Detering KM, Hancock AD, Reade MC, Silvester W. The impact of advance care planning on end of life care in elderly patients: randomised controlled trial. BMJ. 2010 Mar 23;340:c1345. doi: 10.1136/bmj.c1345. PMID 20332506
- [Background] Garrouste-Orgeas M, Tabah A, Vesin A, Philippart F, Kpodji A, Bruel C, Gregoire C, Max A, Timsit JF, Misset B. The ETHICA study (part II): simulation study of determinants and variability of ICU physician decisions in patients aged 80 or over. Intensive Care Med. 2013 Sep;39(9):1574-83. doi: 10.1007/s00134-013-2977-x. Epub 2013 Jun 14. PMID 23765237
- [Derived] Denis N, Timsit JF, Giaj Levra M, Sakhri L, Duruisseaux M, Schwebel C, Merle P, Pinsolle J, Ferrer L, Moro-Sibilot D, Toffart AC. Impact of systematic advanced care planning in lung cancer patients: A prospective study. Respir Med Res. 2020 Mar;77:11-17. doi: 10.1016/j.resmer.2019.09.003. Epub 2019 Oct 28. PMID 31927479